CLINICAL TRIAL: NCT04051710
Title: Randomized, Double Blind, Placebo Controlled, Parallel Group Study to Evaluate Efficacy and Safety of Beclomethasone Dipropionate Metered Dose Inhaler (Inhalation Aerosol) (0.04mg/ INH) in Male and/ or Female Subjects With Asthma
Brief Title: Clinical Pharmacodynamic Bioequivalence Study of Beclomethasone Dipropionate 40 mcg INH
Acronym: QVR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aurobindo Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR176-17
Record Dates: First submitted 2019-08-05; First posted 2019-08-09 (Actual); Results first posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group-I (Test) (Experimental): One inhalation of Beclomethasone dipropionate HFA, 0.04 mg/ INH (Test) twice daily.
  Interventions: Drug: Test Product
- Group-II (Reference) (Active Comparator): One inhalation of QVAR® 40 mcg (Beclomethasone dipropionate HFA), Inhalation Aerosol twice daily.
  Interventions: Drug: Reference Product
- Group-III (Placebo) (Placebo Comparator): One inhalation of Placebo Inhalation Aerosol twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Test Product — Beclomethasone Dipropionate Inhalation Aerosol, 40 mcg
  Other Names: Test
  Arms: Group-I (Test)
Drug: Reference Product — Beclomethasone Dipropionate Inhalation Aerosol, 40 mcg
  Other Names: QVAR
  Arms: Group-II (Reference)
Drug: Placebo — Placebo Product
  Arms: Group-III (Placebo)

SUMMARY:
To compare the therapeutic equivalence of Beclomethasone Dipropionate MDI (Inhalation Aerosol) 0.04 mg/ INH with the marketed QVAR® 40 mcg (Beclomethasone dipropionate hydrofluoroalkane (HFA)) and to demonstrate superiority of both active treatments over placebo.

DETAILED DESCRIPTION:
This study is to demonstrate the pharmacodynamic bioequivalence of the test product to the reference product in terms of improvement in FEV1 measured before and after 4 weeks of treatment in adult patients with chronic stable asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female subjects of non-childbearing or of childbearing potential committing to consistent and correct use of an acceptable method of birth control.
2. Diagnosis of asthma as defined by the National Asthma Education and Prevention Program at least 12 months prior to screening.
3. Pre-bronchodilator FEV1 of >45% and <85% of predicted value during the screening visit and on the first day of treatment.
4. >15% and >0.20 L reversibility of FEV1 within 30 minutes following 360 mcg of albuterol inhalation (pMDI).
5. Patients should be stable on their chronic asthma treatment regimen for at least four weeks prior to enrollment.
6. Currently non-smoking; had not used tobacco products (i.e., cigarettes, cigars, pipe tobacco) within the past year, and having had <10 pack-years of historical use.
7. Ability to replace current short-acting β agonist (SABAs) with salbutamol/albuterol inhaler for use as needed for the duration of the study. Subjects should be able to withhold all inhaled SABAs for at least six hours prior to lung function assessments on study visits.
8. Ability to discontinue their asthma medications (inhaled corticosteroids and long-acting β agonists) during the run-in period and for remainder of the study.
9. Willingness to give their written informed consent to participate in the study.

Exclusion Criteria:

1. Life-threatening asthma, defined as a history of asthma episodes(s) requiring intubation, and/or associated with hypercapnia, respiratory arrest or hypoxic seizures, asthma related syncopal episode(s), or hospitalizations within the past year prior to the screening or during the run-in period.
2. Significant respiratory disease other than asthma (COPD, interstitial lung disease, etc.)
3. Evidence or history of clinically significant disease or abnormality including congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, myocardial infarction, or cardiac dysrhythmia. In addition, historical or current evidence of significant hematologic, hepatic, neurologic, psychiatric, renal, or other diseases that, in the opinion of the investigator, would put the patient at risk through study participation, or would affect the study analyses if the disease exacerbates during the study.
4. Viral or bacterial, upper or lower respiratory tract infection, or sinus, or middle ear infection within four weeks prior to the screening, during the run-in period, or on the day of treatment.
5. Hypersensitivity to any sympathomimetic drug (e.g., albuterol) or any inhaled, intranasal, or systemic corticosteroid therapy.
6. Patients receiving β2-blockers, anti-arrhythmics, anti-depressants, and monoamine oxidase inhibitors within 4 weeks prior to the screening.
7. Patients who required systemic corticosteroids (for any reason) within the past 2 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1550 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Marialouis, Study Director — Aurobindo Pharma USA Inc
Locations (1):
- Maharashtra Medical Foundation Joshi Hospital, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No
Not decided

RESULTS

PARTICIPANT FLOW:
Groups:
- Group I (Test): One inhalation of Beclomethasone dipropionate HFA, 0.04 mg/ INH (Test) twice daily.
  Test Product: Beclomethasone Dipropionate Inhalation Aerosol, 40 mcg
- Group II: One inhalation of Beclomethasone dipropionate HFA, 0.04 mg/ INH (Reference) twice daily.
  Reference Product: QVAR® Beclomethasone Dipropionate Inhalation Aerosol, 40 mcg
- Group III (Placebo): One inhalation of Placebo inhalation aerosol twice daily.
Period: Overall Study
Arm/Group | Group I (Test) | Group II | Group III (Placebo)
Started | 620 | 620 | 310
Completed | 616 | 612 | 306
Not Completed | 4 | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Test Group: Subjects randomly enrolled into test group received test comparator, Beclomethasone dipropinate, 0.04 mg/INH to administer one inhalation twice daily
- Reference Group: Subjects randomly enrolled into Reference group received Reference comparator, QVAR® containing Beclomethasone dipropinate, 0.04 mg/INH to administer one inhalation twice daily
- Placebo Group: Subjects randomly enrolled into Placebo group received a Placebo device to administer one inhalation twice daily
- Total: Total of all reporting groups
Arm/Group | Test Group | Reference Group | Placebo Group | Total
Number analyzed (Participants) | 617 | 615 | 308 | 1540
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (12.71) | 41.8 (12.85) | 40.6 (12.86) | 41.2 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 267 | 272 | 139 | 678
  Male | 350 | 343 | 169 | 862
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 617 | 615 | 308 | 1540
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 617 | 615 | 308 | 1540

OUTCOME MEASURES:

1. Primary Outcome: Change in FEV1 From Pre Dose to End of Treatment
Description: Mean change in Forced Expiratory volume in 1 second (FEV 1) from baseline to end of study visit
Time Frame: 4 weeks
Population: Mean change of FEV1 from baseline to end of study was measured
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Group-I (Test) | Group-II (Reference) | Group-III (Placebo)
Number analyzed (Participants) | 577 | 566 | 282
Litres | 0.23 (0.01) | 0.22 (0.01) | 0.09 (0.01)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Group II (Reference): One inhalation of Beclomethasone dipropionate HFA, 0.04 mg/ INH (Reference) twice daily.
  Reference Product: QVAR® Beclomethasone Dipropionate Inhalation Aerosol, 40 mcg
Arm/Group | Group I (Test) | Group II (Reference) | Group III (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/619 | 0/620 | 0/310
Serious Adverse Events (participants affected / at risk) | 0/619 | 0/620 | 0/310
Other Adverse Events (participants affected / at risk) | 39/619 | 25/620 | 18/310
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group I (Test) (N=619) | Group II (Reference) (N=620) | Group III (Placebo) (N=310)
Headache (Nervous system disorders) | 13 | 7 | 4 — Headache
Tremor (Nervous system disorders) | 0 | 1 | 0
Vertigo (Nervous system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 7 | 5 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 0
Pain (General disorders) | 3 | 0 | 1
Pyrexia (General disorders) | 5 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Migraine (Vascular disorders) | 1 | 0 | 0
Alanine Aminotransferase increased (Investigations) | 1 | 1 | 1
Aspartate Aminotransferase increased (Investigations) | 1 | 1 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0 | 1
white blood cells decreased (Investigations) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the ownership of all the data generated from the study and PI has no rights to publish the results or any information derived from the study.

DOCUMENTS (2):
  • Study Protocol (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT04051710/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT04051710/SAP_001.pdf